CLINICAL TRIAL: NCT02454192
Title: A Study of the Feasibility and Effectiveness of Implementing and Diffusing an Evidence-based Childhood Asthma Management Intervention in Community Health Centers
Brief Title: Community Healthcare for Asthma Management and Prevention of Symptoms
Acronym: CHAMPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Rho, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 31993
Record Dates: First submitted 2015-04-29; First posted 2015-05-27 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Asthma
Keywords: Evidence-based intervention; Implementation; Underserved communities
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHAMPS Intervention (Other): Tailored asthma education and counseling for children with moderate to severe asthma who have confirmed allergies to environmental triggers present in their homes provided through a combination of clinic and home visits
  Interventions: Behavioral: CHAMPS
- Usual Care (No Intervention): Usual asthma care and management

INTERVENTIONS:
Behavioral: CHAMPS
  Arms: CHAMPS Intervention

SUMMARY:
The purpose of this study is to systematically investigate across health center study sites participating in this study the process of adopting, integrating, implementing, and diffusing a minimum set of evidence-based interventions for the management of childhood asthma. Investigators hypothesized that an intervention that is evidence- and consensus-based (i.e., minimum elements to be integrated into existing practice, dosing of each element) would be implemented effectively, as measured by health center performance improvement on child health outcomes, health care utilization, and other measures (e.g., avoidable costs).

DETAILED DESCRIPTION:
In this study, investigators combined childhood asthma counseling and environmental interventions proven effective in previous NIH-funded clinical trials, the National Cooperative Inner-City Asthma Study (NCICAS) and the Inner-City Asthma Study (ICAS), and a third study, Head-off Environmental Asthma in Louisiana (HEAL). These studies demonstrated that participant-tailored interventions reduce asthma morbidity. Through a process of consensus building, investigators adapted a hybrid of these interventions for use in primary care clinics located in medically underserved areas (FQHCs). Investigators recruited participants ages 5-12 years with poorly controlled, moderate-to-severe asthma to ensure comparability with previous studies. Unlike the earlier clinical trials, which limited eligibility to inner-city children in stable housing, CHAMPS enrolled participants regardless of housing situation (e.g., temporary/shared homes) and location (e.g., urban/rural). Investigators collaborated with 3 FQHCs in Arizona, Michigan, and Porto Rico to enroll children and implement the CHAMPS intervention but otherwise granted them discretion to make decisions about staffing, patient flow and other process determinations, while tracking what those entailed. Investigators also invited 3 additional FQHCs to recruit and enroll children in a comparison group that did not receive the intervention.

The primary aim is to identify and understand barriers and solutions to the adaptation of an evidence-based asthma intervention at the system-level. The evaluation consists of determining how a system makes room for an intervention, identifying stakeholders to make it happen, documenting the process for replication, and monitoring processes and outcomes to ensure the integrity of the intervention remains intact. The process of implementation in the unique clinical settings presented by health centers will be described, including the facilitators and the barriers to the systematic adoption of an evidence-based childhood asthma intervention into routine practice. Of particular importance are those determinants related to in-home and community-based environmental risks, the limits of understanding on the part of parents and caretakers, and community-wide policies and practices that may create health risks.

The secondary aim is to assess the effectiveness and cost-effectiveness of the evidence-based asthma intervention as implemented in health centers.

The third and final aim is to develop a dissemination strategy and some tools for further take up of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma
* Currently receiving long-term asthma control therapy and either has symptoms consistent with persistent asthma or has evidence of uncontrolled disease or is not currently receiving long-term asthma control therapy and has symptoms consistent with persistent asthma and also has evidence of uncontrolled disease
* Caretaker speaks English or Spanish

Exclusion Criteria:

* Younger or older children
* Mild, intermittent asthma

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 599 (Actual)
Dates: Start 2010-10; Primary Completion 2015-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Asthma symptoms | In the past 4 weeks
  Reduction in asthma symptom days in the past 4 weeks as measured by the Asthma Symptoms and Utilization (ASU) questionnaire

SECONDARY OUTCOMES:
Utilization of health care services | In the past year
  Reduction of utilization of Emergency Departments and hospitalizations in the past 12 months as measured by the Asthma Symptom and Utilization (ASU) questionnaire

OTHER OUTCOMES:
Success of implementation | 5 years
  Successful implementation of the CHAMPS intervention at health centers during the study period as measured by different aspects of implementation (see Outcomes 4-9) as measured by different instruments, including fidelity index, ASU, modified CAHPS and attitude patient surveys, provider interviews, leadership interviews, and Medicaid health plan claims data
Success of implementation | 5 years
  Successful implementation of the CHAMPS intervention at health centers during the study period as measured by close fidelity to intervention protocol as measured by fidelity index
Success of implementation | 5 years
  Successful implementation of the CHAMPS intervention at health centers during the study period as measured by improvement in clinical outcomes (i.e., reduction in asthma symptom days) as measured by ASU
Success of implementation | 5 years
  Successful implementation of the CHAMPS intervention at health centers during the study period as measured by high satisfaction/change in attitudes about home visits among caretakers as measured by modified Consumer Assessment of Healthcare Providers and Systems (CAHPS) and patient attitude surveys
Success of implementation | 5 years
  Successful implementation of the CHAMPS intervention at health centers during the study period as measured by change in providers' perceptions of benefit of CHAMPS as measured by provider interviews
Success of implementation | 5 years
  Successful implementation of the CHAMPS intervention at health centers during the study period as measured by leadership intent to sustain services included in CHAMPS as measured by leadership interviews
Success of implementation | 5 years
  Successful implementation of the CHAMPS intervention at health centers during the study period as measured by decrease in costs, especially among high users, as measured by ASU questionnaire and Medicaid health plan claims data

CONTACTS AND LOCATIONS:
Overall Officials: Anne R Markus, JD, PhD, MHS, Principal Investigator — George Washington University; Herman Mitchell, PhD, Principal Investigator — Rho, Inc.
Locations (1):
- Milken Institute School of Public Health, Washington D.C., District of Columbia, United States